CLINICAL TRIAL: NCT00584116
Title: Balloon Aortic Valvuloplasty During Surgical Aortic Valve Replacement
Acronym: BAV-SAVR
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200614760
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Aortic Stenosis
Keywords: Aortic Valve Replacement; AVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prospective, two academic center, non-randomized pilot, acute in-patient study correlating pre-operative imaging studies, intra-operative measurements and intra-operative balloon aortic valvuloplasty (BAV) in patients with degenerative aortic stenosis undergoing surgical aortic valve replacement (SAVR) to understand the requirements (device size and radial strength) of emerging percutaneous heart valve technologies in the treatment of aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Any patient with severe, symptomatic calcific aortic stenosis (AS) referred for elective surgical aortic valve replacement.

  * Severe AS: aortic valve area (AVA) ≤ 1.0 cm2
  * Symptoms: dyspnea on exertion, heart failure, angina or syncope believed to be secondary to AS

Exclusion Criteria:

* Emergent surgical aortic valve replacement.
* Inability to undergo TTE or TEE intra-operatively.
* Currently participating in another study that has not completed the primary endpoint or that clinically interferes with the current study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with severe symptomatic calcific aortic stenosis (AS) referred for elective surgical aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
aortic annulus size | 2 months
  Show the correlation between the size of the aortic annulus measured intra-operatively with surgical rings (gold standard) with other methods of aortic annulus measurement that would not require surgical intervention (CT, TEE, TTE)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Rogers, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- See also: Clinical Trials at UC Davis Medical Center — http://www.ucdmc.ucdavis.edu/clinicaltrials/